CLINICAL TRIAL: NCT07227857
Title: A Phase Ib/II First-in-human, Multicentre, Open-label, Multiple Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamic Effect of Intrathecal S230815 in Pediatric Participants With KCNT1-related Developmental and Epileptic Encephalopathy
Brief Title: A First-in-human Study of S230815 in Pediatric Participants With KCNT1-related Developmental and Epileptic Encephalopathy
Acronym: KANDLE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CL1-230815-001; 2024-513332-17-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-12; First posted 2025-11-13 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Epileptic Encephalopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental)
  Interventions: Drug: S230815- Starting dose A
- Cohort 2 (Experimental)
  Interventions: Drug: S230815- Dose B
- Cohort 3 (Experimental)
  Interventions: Drug: S230815- Dose C
- Cohort 4 (Experimental)
  Interventions: Drug: S230815- Dose D

INTERVENTIONS:
Drug: S230815- Starting dose A — Solution for injection
  Arms: Cohort 1
Drug: S230815- Dose B — Solution for injection
  Arms: Cohort 2
Drug: S230815- Dose C — Solution for injection
  Arms: Cohort 3
Drug: S230815- Dose D — Solution for injection
  Arms: Cohort 4

SUMMARY:
Study CL1-230815-001 (KANDLE) is a Phase Ib/II, First In Human, multicentre, open-label, multiple ascending dose study to assess the safety, tolerability, pharmacokinetics (PK) and pharmacodynamic (PD) effect of S230815 in pediatric participants with KCNT1-related Developmental Epileptic Encephalopathy. To participate in the study, participants must have a diagnosis of Developmental Epileptic Encephalopathy due to a documented pathogenic or likely pathogenic variant in KCNT1 (to be confirmed by central genetic testing at the screening visit). The study consists of a screening period followed by two consecutive interventional parts. Part 1 will evaluate multiple ascending doses of S230815. Part 2 is a long-term treatment extension for participants who have completed Part 1. Participants will seamlessly roll-over from Part 1 to Part 2, resuming the same cohort as they were assigned in Part 1, and will receive S230815 for a maximum of 72 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female pediatric participants aged 2-12 years old at screening, with a genetically confirmed diagnosis of Developmental Epileptic Encephalopathy (DEE) due to a pathogenic or likely pathogenic variant in KCNT1 confirmed by central genetic testing.
* Stable dose of other regular medications and/or stable antiseizure interventions (such as ketogenic diet and vagal nerve stimulation).

Exclusion Criteria:

* Other clinical phenotypes associated with pathogenic or likely pathogenic variants in KCNT1 other than Epilepsy of Infancy with Migrating Focal Seizures or Early-Onset Epileptic Encephalopathy
* Documented pathogenic or likely pathogenic variants in any other gene known to cause epilepsy identified through prior genetic testing. Variants of uncertain significance in other genes known to cause epilepsy may be considered on discussion with the sponsor.
* Clinically significant medical history or clinical findings on physical examination, other than DEE, that in the judgment of the investigator, make the participant unsuitable for participation in the study and/or completion of the trial procedures, including, but not limited to:

  * Clinically significant prior or ongoing medical conditions within 30 days of the screening visit, as per investigator judgement.
  * Clinically significant abnormality on Electrocardiogram (ECG) at the screening visit, as per investigator judgement.
  * Clinically significant abnormality on laboratory testing at screening, including, but not limited to:
  * Renal insufficiency, which is defined as creatinine clearance < 40 mL/min assessed as estimated glomerular filtration rate (eGFR) using Modification of Diet in Renal Disease (MDRD) formula
  * Hepatic derangement defined as transaminase values more than 3 times the Upper Limit of Normal (ULN) range, or total bilirubin values more than 1.5 times the ULN.
* Positive hepatitis B surface antigen test, positive hepatitis C antibody test, positive for human immunodeficiency virus (HIV), as reported by a laboratory test within 6 months prior to the screening visit, or on screening bloods.
* Bone, spine, bleeding disorders, or other disorder that exposes the participant to risk of injury or unsuccessful Lumbar puncture (e.g., haemophilia, Von Willebrand's disease, liver disease).
* Contraindications to undergoing Magnetic Resonance Imaging (MRI), Lumbar puncture procedure and Intrathecal administration.
* History of Central Nervous System (CNS) tumors or malignancies, including CNS metastatic disease.
* Continuous respiratory support, defined as oxygen supplementation or non-invasive ventilation (e.g.: continuous positive airway pressure, bi-level intermittent positive airway pressure), required during waking hours. This does not include suctioning; cough assist devices or other devices that may be used regularly to clear airways.
* Invasive ventilation including the presence of a tracheostomy.
* Use of quinidine within 30 days prior to the screening visit.
* Current use or anticipated use of antiplatelet or anticoagulant therapy during the study.
* Current or past enrolment in an interventional clinical study in which an investigational therapy is/was administered within 30 days (or 5 half-lives of study agent, whichever is longer) prior to the screening visit.
* Implantable CNS device that may interfere with the ability to administer the study drug via Lumbar puncture.
* Known hypersensitivity to any oligonucleotide, as demonstrated by a systemic allergic reaction (e.g., changes in pulse, blood pressure, breathing function, etc.), or any other drug that in the opinion of the investigator may preclude study participation.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2028-04-15 (Estimated); Study Completion 2028-04-15 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of Adverse Events (AE)'s. | Through End of study visit (A maximum of 116 weeks)

SECONDARY OUTCOMES:
Pharmacokinetic (PK) parameters of S230815 in cerebrospinal fluid (CSF) Ctrough | Through week 96
  Ctrough is defined as the concentration reached immediately before the next dose is administered.
Pharmacokinetic (PK) parameters of S230815 in plasma AUC 0-τ | Through End of study visit (A maximum of 116 weeks)
  Area Under the Curve (AUC) from dosing (time 0) to time t [AUC0-t]
Pharmacokinetic (PK) parameters of S230815 in plasma Cmax | Through End of study visit (A maximum of 116 weeks)
  Cmax is defined as the maximum (peak) observed concentration following a dose. Measured 0.5, 2, 4, 8 , and 24 hours post dose
Pharmacokinetic (PK) parameters of S230815 in plasma Ctrough | Through End of study visit (A maximum of 116 weeks)
Relative change from baseline in seizure frequency as recorded by daily seizure logs | Through End of study visit (A maximum of 116 weeks)
Relative change from baseline in seizure frequency as recorded by periodic 24h Video Electroencephalogram (vEEG) assessment | Through End of study visit (A maximum of 116 weeks)
Number and administration frequency of rescue medication | Through End of study visit (A maximum of 116 weeks)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (6):
  - Children's Hospital of Orange County, Orange, California
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Rochester Medical Center, Rochester, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Health Dallas, Dallas, Texas
- France (3):
  - Institut Des Neurosciences De La Timone, Marseille
  - Hopital Necker Enfants Malades, Paris
  - Robert Debre University Hospital, Paris
- Italy (2):
  - Azienda Ospedaliera Universitaria Meyer IRCCS, Florence
  - Ospedale Pediatrico Bambino Gesu, Roma
- Japan (3):
  - Shinshu University Hospital, Nagano
  - Osaka City General Hospital, Osaka
  - Shizuoka Institute of Epilepsy and Neurological Disorders, Shizuoka
- Spain (2):
  - Hospital Sant Joan De Deu Barcelona, Esplugues de Llobregat
  - Hospital Ruber Internacional, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.